CLINICAL TRIAL: NCT02076386
Title: A Prospective, Non-interventional Study of the Use of Dolutegravir as Part of Combination Antiretroviral Therapy in Routine Daily Practice in Germany (DOL-ART)
Brief Title: A Prospective, Non-interventional Study of the Use of Dolutegravir as Part of Combination Antiretroviral Therapy in Routine Daily Practice in Germany
Acronym: DOL-ART
Status: Completed | Type: Observational
Sponsor: ViiV Healthcare (Industry)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 201067
Record Dates: First submitted 2014-02-20; First posted 2014-03-03 (Estimated); Last update posted 2018-08-13 (Actual); Status verified 2018-08

CONDITIONS: Infection, Human Immunodeficiency Virus
MeSH Terms: conditions — Infections; Acquired Immunodeficiency Syndrome | interventions — dolutegravir

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Dolutegravir: Prospective, non-interventional study of the use of doluetegravir as part of an antiretroviral combination therapy in routine daily practice in Germany. No drug will be provided. No study visits or procedures are mandated per protocol.
  Interventions: Drug: Dolutegravir

INTERVENTIONS:
Drug: Dolutegravir — Prospective, non-interventional study of the use of doluetegravir as part of an antiretroviral combination therapy in routine daily practice in Germany. No drug will be provided. No study visits or procedures are mandated per protocol.

SUMMARY:
DOL-ART is a multi-center, prospective, non-interventional study of the use of doluetegravir as part of an antiretroviral combination therapy in routine daily practice in Germany. The primary study objective is a descriptive characterization of the frequency of therapeutic monitoring measures in HIV-infected patients under dolutegravir-containing ART in routine daily practice in Germany.

The study is designed to enroll approximately 400 patients. There are no protocol-mandated visits or procedures associated with the study. Each patient is expected to participate for a maximum of 3 years or until premature discontinuation (i.e., discontinuation of dolutegravir, due to death, withdrawal of consent, lost to follow-up).

ELIGIBILITY:
Inclusion Criteria:

* Documented HIV infection
* Age ≥ 18 years
* Decision for the first initiation of dolutegravir as part of an ART by the attending physician irrespective of inclusion in this observational study
* Prior to the start of this study, the patient must have been receiving a dolutegravir-containing ART for at least 4 weeks

Exclusion Criteria:

* Discontinuation of dolutegravir as part of an ART prior to the start of the study documentation
* Participation in a clinical trial during this study
* Participation in a clinical trial or compassionate use program with dolutegravir being or having been part of the investigational medication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Approximately 40 HIV treatment centers in Germany are planned to be involved in the documentation. The participating study site will document a maximum of 20 patients for this observation study. Overall, approximately 400 patients under dolutegravir-containing ART are to be documented. This selection process is intended to achieve the documentation of patients under dolutegravir-containing ART in routine daily practice representative for Germany.
Sampling Method: Non-Probability Sample
Enrollment: 411 (Actual)
Dates: Start 2014-03-04 (Actual); Primary Completion 2017-07-05 (Actual); Study Completion 2017-07-05 (Actual)

PRIMARY OUTCOMES:
Frequency of therapeutic monitoring measures in HIV-infected patients | up to 3 years
  Descriptive characterization of the frequency of therapeutic monitoring measures in HIV-infected patients under dolutegravir-containing ART in routine daily practice in Germany.

SECONDARY OUTCOMES:
Type of the therapeutic monitoring measures | up to 3 years
Number of participants with Serious Adverse Events and drug-related adverse events as a measure of safety and tolerability | up to 3 years
  To evaluate the frequency and type of serious adverse events and drug-related adverse events in patients treated with dolutegravir.
Efficacy | from start of dolutegravir up to 3 years
  Defined as viral load < 50 copies/ml
Resistance profile | from start of dolutegravir up to 3 years
  To characterise resistance profile in case of virological failure
Patient satisfaction | Up to 3 years from baseline
  To evaluate the change in patient satisfaction relative to baseline in patients treated with dolutegravir
Reasons for selecting dolutegravir-containing ART | Baseline
Reasons for discontinuing dolutegravir-containing ART | Up to 3 years after baseline

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — ViiV Healthcare
Locations (23):
- Germany (23):
  - GSK Investigational Site, Freiburg im Breisgau, Baden-Wurttemberg
  - GSK Investigational Site, Mannheim, Baden-Wurttemberg
  - GSK Investigational Site, Stuttgart, Baden-Wurttemberg
  - GSK Investigational Site, Tübingen, Baden-Wurttemberg
  - GSK Investigational Site, Fürth, Bavaria
  - GSK Investigational Site, Munich, Bavaria
  - GSK Investigational Site, Frankfurt am Main, Hesse
  - GSK Investigational Site, Hanover, Lower Saxony
  - GSK Investigational Site, Osnabrück, Lower Saxony
  - GSK Investigational Site, Aachen, North Rhine-Westphalia
  - GSK Investigational Site, Bochum, North Rhine-Westphalia
  - GSK Investigational Site, Cologne, North Rhine-Westphalia
  - GSK Investigational Site, Dortmund, North Rhine-Westphalia
  - GSK Investigational Site, Düsseldorf, North Rhine-Westphalia
  - GSK Investigational Site, Münster, North Rhine-Westphalia
  - GSK Investigational Site, Koblenz, Rhineland-Palatinate
  - GSK Investigational Site, Mainz, Rhineland-Palatinate
  - GSK Investigational Site, Magdeburg, Saxony-Anhalt
  - GSK Investigational Site, Berlin
  - GSK Investigational Site, Chemnitz
  - GSK Investigational Site, Cologne
  - GSK Investigational Site, Hamburg
  - GSK Investigational Site, Weimar